CLINICAL TRIAL: NCT03473704
Title: Assessment of the Effectiveness of a New Telematic Program for the Treatment of Depression in Patients With Type 1 Diabetes
Brief Title: Telematic Program for the Treatment of Depression in Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: University of Malaga (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WEB_TDDI1 STUDY
Record Dates: First submitted 2018-03-06; First posted 2018-03-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Type 1 Diabetes Mellitus; Depression
Keywords: Type 1 diabetes; Depression; Telematic Program; Treatment; Web-based
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Depression | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The treatment group (TG) will receive the web treatment, which consists of 9 weekly sessions, while the control group (CG) will be evaluated in the same phases as the TG. For ethical reasons, the CG will receive the web treatment once the TG intervention has been completed. There will be a follow-up at 3, 6 and 12 months.
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (TG) (Experimental): The treatment group (TG) will receive the web treatment, which consists of 9 weekly sessions.
  Interventions: Behavioral: Treatment group (TG)
- Control group (CG) (Placebo Comparator): The control group (CG) will be evaluated in the same phases as the TG.
  Interventions: Behavioral: Control group (CG)

INTERVENTIONS:
Behavioral: Treatment group (TG) — The Treatment group (TG) will receive the web treatment, which consists of 9 weekly sessions.
  Arms: Treatment group (TG)
Behavioral: Control group (CG) — For ethical reasons, the CG will receive the web treatment once the TG intervention has been completed (as long as it continues to meet the conditions of the study).
  Arms: Control group (CG)

SUMMARY:
In diabetes, web programs have been designed that have integrated cognitive-behavioral therapy (CBT) with diabetes education, obtaining positive results in the mood of the patient. In Spain, no similar approach has been performed in people with diabetes and depression. However, the need to provide professionals with adequate tools to help people with this problem is justified.

The main objective of this project is to apply a telematic program for the treatment of specific depression for people with type 1 diabetes designed by our research team in a sample of patients with type 1 diabetes and mild-moderate depressive symptomatology of the province of Malaga. To do this, the sample will be divided into two groups: treatment group (TG) and control group (CG). The design of the study is quasi-experimental, longitudinal randomized pre-post with control group. The treatment group (TG) will receive the web treatment, which consists of 9 weekly sessions, while the control group (CG) will be evaluated in the same phases as the TG. For ethical reasons, the CG will receive the web treatment once the TG intervention has been completed. There will be a follow-up at 3, 6 and 12 months.

DETAILED DESCRIPTION:
On the website will be collected the 9 sessions of which the treatment consists. The sessions will be weekly. Each week, the patient will find a brief summary of the previous session and an introduction to the topic, where the new session will be explained. Then, the patient will be provided with the new information (the topic treated) and different examples will be added to facilitate understanding. Once the information is presented, a summary of the key ideas of the session and a small evaluation to assess the understanding on the part of the patient will be presented. At the end of the session, the patient will have the key ideas and a self-evaluation of the session. Finally, the patient will be explained the task to be performed and sent to the therapist with an example of how to perform it. In addition, the patient will have a bibliography of each of the topics discussed. Each session will last 20-30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Have a medical diagnosis of type 1 diabetes ≥1 year;
* be over 18 years old;
* have a psychological diagnosis of mild / moderate major depressive disorder, dysthymia or depressive symptomatology;
* not have a concomitant pharmacological treatment that could modify the glycaemia values or the depressive symptomatology;
* not be in previous psychological treatment;
* absence of:
* chronic renal failure,
* impaired liver function tests,
* active thyroid disease (except correctly substituted hypothyroidism),
* gestation in progress;
* absence of acute ketosis decompensation at the beginning of the study;
* have access to the internet.

Exclusion Criteria:

* Type 2 diabetes;
* pregnant women or planning pregnancy;
* severe macro or microvascular complications;
* diagnosis of severe major depressive disorder with suicide risk;
* no collaboration (no informed consent signature);
* not have access to the internet;
* present a disabling psychiatric disorder, psychosis, diagnosis of severe depressive disorder, suicidal ideation;
* not have access to the internet.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-19 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Depression | Change between Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-5 (SCID-5)
Depression symptoms | Change between Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Beck Depression Inventory-Fast Screen (BDI-FS)

SECONDARY OUTCOMES:
Fear of Hypoglycemia | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Fear of Hypoglycemia Scale (FH-15): 15 summable items assessed on a 5-point Likert scale with a range of 1-5. The cutoff score was set at 28 points. Individuals with scores equal to or greater than 28 points will be classified as having fear of hypoglycemia.
Distress | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Diabetes Distress Scale (DDS): 17 items measure that uses a Likert scale to score each item from 1 (no problem) to 6 (a serious problem) during the last month. Based on four distress-related domains: emotional burden subscale, physician-related distress subscale, regimen-related distress subscale, and diabetes-related interpersonal distress.
Quality of Life | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Diabetes Quality of Life Questionnaire (DQOL)
Anxiety | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  The State-Trait Anxiety Inventory (STAI)
Coping | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Coping Inventory (COPE)
Personality | Pre treatment.
  Millon Clinical Multiaxial Inventory (MCMI-III)
Adherence | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Self-Care Inventory-revised (SCI-R)
Glycemic control | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Glycosylated hemoglobin test (HbA1c)
Hypoglycemia | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Number of mild hypoglycemia weekly and severe hypoglycaemia in the last year.
Hyperglycemia | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Number of hyperglycemia weekly.
Ketone | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Number of ketone test positive in the last year.
Blood glucose self-tests | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Number of blood glucose self-tests daily.
Complications of diabetes | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Collect if there is any complication of diabetes in the patient's clinical history.
Another disease | Pre treatment, post treatment (12 weeks), 3, 6 and 12 months.
  Collect if there is any illness (other than diabetes) diagnosed by the doctor in the patient's clinical history.

CONTACTS AND LOCATIONS:
Overall Officials: María Teresa Anarte, PhD, Principal Investigator — University of Malaga
Locations (1):
- University of Malaga, Málaga, Spain

REFERENCES:
- [Background] van Bastelaar KM, Pouwer F, Cuijpers P, Twisk JW, Snoek FJ. Web-based cognitive behavioural therapy (W-CBT) for diabetes patients with co-morbid depression: design of a randomised controlled trial. BMC Psychiatry. 2008 Feb 19;8:9. doi: 10.1186/1471-244X-8-9. PMID 18284670
- [Background] van der Feltz-Cornelis CM, Nuyen J, Stoop C, Chan J, Jacobson AM, Katon W, Snoek F, Sartorius N. Effect of interventions for major depressive disorder and significant depressive symptoms in patients with diabetes mellitus: a systematic review and meta-analysis. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):380-95. doi: 10.1016/j.genhosppsych.2010.03.011. Epub 2010 May 15. PMID 20633742
- [Derived] Carreira M, Ruiz de Adana MS, Pinzon JL, Anarte-Ortiz MT. Internet-based cognitive-behavioral therapy is effective in reducing depressive symptomatology in type 1 diabetes: results of a randomized controlled trial. Front Clin Diabetes Healthc. 2023 Nov 7;4:1209236. doi: 10.3389/fcdhc.2023.1209236. eCollection 2023. PMID 38028977
- [Derived] Carreira M, Ruiz de Adana MS, Pinzon JL, Anarte-Ortiz MT. Internet-based Cognitive-behavioral therapy (CBT) for depressive symptomatology in individuals with type 1 diabetes (WEB_TDDI1 study): A randomized controlled trial protocol. PLoS One. 2022 Sep 20;17(9):e0274551. doi: 10.1371/journal.pone.0274551. eCollection 2022. PMID 36126050